CLINICAL TRIAL: NCT04257422
Title: Intentional Rounding in Internal Medicine: a Multicenter, Randomized National Study Studio INTENTO - FADOI.03.2018
Brief Title: Intentional Rounding in Internal Medicine
Acronym: INTENTO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrolment for the study ended concurrently with the development of the CoViD-19 pandemic. This decision was made by the Steering Committee in consideration of the transformation of some wards participating in the study into CoVID-19 units.
Sponsor: Fadoi Foundation, Italy (Other)
Collaborators: ANìMO (Associazione Nazionale Infermieri Medicina) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FADOI.03.2018
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hospitalization
Keywords: Nursing

STUDY DESIGN:
Intervention Model Description: Cluster randomized
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intentional Rounding (Experimental): In the centers randomized to Intentional Rounding the ward nurses will have to adopt a new proactive care method towards hospitalized patients
  Interventions: Other: Intentional Rounding
- Control (No Intervention): In randomized controlled centers, nurses guarantee the standard care provided by the ward

INTERVENTIONS:
Other: Intentional Rounding — A new method of nursing care named Intentional Rounding. The "intentional roundings" are planned rounds, conducted at regular intervals by nursing staff to anticipate care, comfort, hospitality and psychological needs of hospitalized users.
  Arms: Intentional Rounding

SUMMARY:
Each investigator will have to collect data for 50 hospitalized patients in the Internal Medicine wards. If the center is randomized to Intentional Rounding, the staff of nurses and OSS will have to implement the new care strategy.

DETAILED DESCRIPTION:
The centers participating in the study are randomized to the Intentional Roundig group and the Control group, in a 1: 1 ratio. In the randomized centers for experimental intervention, a training intervention lasting about 4 hours was conducted by a nurse expert in Intentional Rounding.

At the end of the study, training is also scheduled for the Control Centers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signature of informed consent
* Patients who understand Italian

Exclusion Criteria:

* Patients who deny informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1822 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
Falls and new bedsores | 3 months
  Cumulative assessment of the incidence of falls and the appearance of new pressure sores in hospitalized patients in the Internal Medicine wards

SECONDARY OUTCOMES:
Call lights | 3 months
  Analysis of the impact of the implementation of Intentional Rounding on the call lights by hospitalized patients.
  The total number of calls to the emergency bell is evaluated. A call light log will be used on which the nurses will report the reason for each call by the patient.
Measurement of patient satisfaction with the nursing care received and hospitalization | 3 months
  Assessment of the relationship between implementation of the Intentional Rounding and level of patient satisfaction, defined on the basis of how patients consider the way care is provided useful, effective and advantageous (for patients able to perform this evaluation).
  The information will be collected through a questionnaire consisting of two questions. The patient will have to evaluate the nursing care and hospitalization, assigning a score from 1 to 7 (where 1 = bad; 7 = excellent).
Critical thinking of nurses | 3 months
  Evaluation of the critical thinking of nurses following the implementation of Intentional Rounding in clinical practice, defined as the process that is used by nurses when they have to make a clinical decision and manage daily problems (on a voluntary basis between the participating Centers).
  Clinical decision making in nursing scale (CDMNS) will be used to evaluate the critical thinking of nurses.
  For each of the 40 statements, the nurse must think about how she would behave during patient care.
  There are no "right" or "wrong" answers. What matters is his evaluation of how he usually acts in making decisions in clinical reality.
  The answers can be:
  * Always: what he constantly does every time.
  * Frequently: what he usually does in most cases.
  * Occasionally: what he does a few times.
  * Rarely: what he seldom does.

CONTACTS AND LOCATIONS:
Overall Officials: Dino Stefano Di Massimo, Principal Investigator — ANìMO
Locations (23):
- Italy (23):
  - Ospedale Civile Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale San Donato, Arezzo
  - Ospedale degli Infermi, Biella
  - Ospedale "Bernardino Ramazzini", Carpi
  - Ospedale di Castelfranco Veneto, Castelfranco Veneto
  - Ospedale Poveri Infermi, Cuneo
  - Presidio Ospedaliero Pubblico " Santa Croce ", Fano
  - AOU Careggi, Florence
  - Policlinico San Martino, Genova
  - Ospedale S. Andrea, Massa Marittima
  - Fondazione Don Gnocchi, Milan
  - Ospedale Civile di Montebelluna, Montebelluna
  - Ospedale Buonconsiglio Fatebenfratelli, Napoli
  - Ospedale di Noventa Vicentina, Noventa Vicentina
  - Ospedale Buccheri La Ferla FBF, Palermo
  - Ospedali Riuniti Villa Sofia, Palermo
  - Ospedale di Rho, Rho
  - Ospedale FBF Isola Tiberina, Roma
  - Ospedale Civile SS. Annunziata, Savigliano
  - Ospedale San Paolo, Savona
  - AOUS, Siena
  - Ospedale Dell'Alta Val D'Elsa, Siena
  - Ospedale San Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No